CLINICAL TRIAL: NCT02251639
Title: Evaluation of Diagnostic Aids for Detection and Diagnosis of Oral Cancer
Brief Title: Diagnostic Aids for Detection and Diagnosis of Oral Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study design improvements.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); William Marsh Rice University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-0887; NCI-2014-02105 (Registry Identifier: NCI CTRP); RO1 910576 (Other Grant/Funding Number: NCI); 960113 (Other Grant/Funding Number: CPRIT)
Record Dates: First submitted 2014-09-23; First posted 2014-09-29 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Head and Neck Cancer
Keywords: Oral cancer; Pre-cancer; Widefield Fluorescence Imaging; VELScope; Point Spectroscopy System; Oral brush biopsy; Questionnaire; Survey; Diagnostic aid; Screening
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Oral Imaging and Cytology (Experimental): Participant completes a short questionnaire regarding their awareness of oral cancer and risk factors. Oral cavity inspected using a standard white light headlamp. Oral cavity then examined with one or more of the widefield imaging devices, such as the VELscope and/or PS2 device. Exfoliative cells for cytology from an abnormal area (if present) and from a contralateral normal appearing area obtained using a brush.
  Interventions: Behavioral: Questionnaire; Device: POS + PS2 + VELscope; Procedure: Oral Brush Biopsy

INTERVENTIONS:
Behavioral: Questionnaire — Participant completes a short questionnaire regarding their awareness of oral cancer and risk factors.
  Other Names: Survey
Device: POS + PS2 + VELscope — Oral cavity examined with one or more of the widefield imaging devices, such as the VELscope and/or PS2 device.
Procedure: Oral Brush Biopsy — If abnormal areas found, a small brush is pressed against an area inside mouth, and turned 5-10 times. The areas that could be biopsied include gums, tongue, roof of mouth, bottom of mouth, or the inside of cheeks.

SUMMARY:
The goal of this clinical study is to find out if certain instruments/devices, such as wide field fluorescence imaging point spectroscopy and/or brush cytology, can help health care providers find mouth cancer more quickly than a standard oral clinical exam.

DETAILED DESCRIPTION:
Study Procedures:

Certain types of light may cause cells to give off a tiny amount of light (called fluorescence). Researchers have learned that cancer cells and normal cells reflect light and give off fluorescence differently. Researchers want to find out if different kinds of light can be used to discover areas of the mouth that may have abnormal or cancerous cells.

If you agree to take part in this study, a researcher may use up to 3 types of imaging instruments to take pictures and readings of several areas in your mouth.

* VELScope is an FDA approved handheld camera device that takes images of the mouth with different colors of light. The VELScope shines blue light into the mouth, and pictures are taken using a camera that is attached to the device.
* Widefield Fluorescence Imaging uses a non-contact imaging device similar to the VELScope. It shines different colors of light and then takes pictures of the inside of the mouth using a digital camera.
* Point Spectroscopy System uses a probe (about the size of a tip of a pen) that is gently placed on several areas of the mouth. Different colors of light are directed through optic fibers to the lining of the mouth, and the probe collects the light that returns from the tissue and sends the information to a computer.

Researchers will record whether the doctors find any areas within your mouth that may not appear completely normal. They will collect tissue samples of these abnormal areas using a brush biopsy. To perform an oral brush biopsy, the research will press a small brush against an area inside your mouth, and turn it 5-10 times. The areas that could be biopsied include your gums, tongue, the roof of your mouth, the bottom of your mouth, or the inside of your cheeks. Any cells collected from the inside of your mouth will be placed on slides to be studied by the study team.

The samples being collected will only be used for this testing, and no leftover samples will be kept by the research staff.

These procedures should take about 20 minutes total.

This is an investigational study. The VELScope is an FDA approved device and is commercially available. Wide-field and point spectroscopy systems are not FDA approved and are only authorized for research. Up to 500 participants will take part in this multicenter study. Up to 250 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 years and older who are willing to participate.
2. Persons presenting for: Physical or dental exams at outside health care centers OR Research meetings/gatherings OR Subjects identified at MDACC who are not already diagnosed with oral cancer or pre oral cancer: this includes patients with malignancies other than oral cancer, and visitors and family members, attendees of the HNS Oral Cancer Screening event who are willing to participate.

Exclusion Criteria:

1. Subjects with a current diagnosis of oral cancer.
2. Subjects under the age of 18. It is extremely unusual for children to develop oral cancer, therefore data from persons younger than 18 may add unexpected variables which could affect data analysis.
3. Subjects who are unable or unwilling to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Performance of the POS, PS2 and VELscope as Diagnostic Aid for Oral Cancer | 1 day
  Information obtained from the fluorescence and reflectance images, point spectroscopy, and oral cytology compared with clinical diagnosis to evaluate the performance of the diagnostic aids and assess any clinical benefit to assist in screening for oral cancer. ROC curve analysis used as primary method for evaluating the performance of the POS, PS2 and VELscope devices as compared to the white light standard clinical diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Gillenwater, MD, BA, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org